CLINICAL TRIAL: NCT05922553
Title: The Effectiveness of Mukbang in Helping Children With Cancer Hospitalized for Radiotherapy and Chemotherapy to Improve Appetite, Nutritional Status and Quality of Life: A Randomized Control Trial
Brief Title: Using Mukbang to Improve Appetite, Nutritional Status and Quality of Life in Children With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wei XIA, PhD (Other)
Responsible Party: Sponsor-Investigator, Wei XIA, PhD, Philosophic Doctor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: mukbang RCT
Record Dates: First submitted 2023-06-05; First posted 2023-06-28 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Children With Cancer
Keywords: Childhood Cancer; Mukbang; Appetite; Nutritional Status; Quality of Life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Ingredient Mukbang (Experimental): Active Ingredient Mukbang will be allocated to the participants in the experimental group. The videos which presented the food images, eating sound and a relaxing and pleasant atmosphere will be sent in sequence through the short video platforms on the smart phone to the participants in the experimental group.
  Interventions: Behavioral: Active Ingredient Mukbang
- General short videos (Placebo Comparator): General short videos without food cues will be allocated to the participants in the placebo control group. There will be no restrictions on the type of short video platforms and specific video content.
  Interventions: Behavioral: General short videos

INTERVENTIONS:
Behavioral: Active Ingredient Mukbang — Mukbang videos include the items which can truly improve the appetite of children with cancer, such as food images, eating sound and interactivity.
  Arms: Active Ingredient Mukbang
Behavioral: General short videos — Short videos that don't contain any food cues.
  Arms: General short videos

SUMMARY:
This study aims to use a two arms randomized clinical trial study to evaluate the effectiveness of the effective constituent of Mukbang in helping children with cancer hospitalized for radiotherapy and chemotherapy to improve their appetite, nutritional status and quality of life.

DETAILED DESCRIPTION:
Cancer has a high incidence among children and adolescents worldwide. In October 2020, the World Health Organization (WHO) released an overview of the Global Action on Childhood Cancer which showed that more than 400,000 children under the age of 19 were diagnosed with cancer worldwide every year. With the development and progress of diagnosis and treatment technology, the health outcome of children with cancer has been greatly improved.

However, the side effects and complications associated with cancer and its treatment can seriously affect the appetite and food intake of children with cancer, resulting in malnutrition and a low quality of life. Therefore, it is very important to effectively improve the appetite of children with cancer during treatment.

Clinical methods to improve the appetite of cancer patients mainly include drugs, diet or nutrition intervention, traditional Chinese medicine and acupuncture, but each intervention has its own advantages and disadvantages which makes the clinical application effect difficult to evaluate, in urgent need of more effective solutions to solve this problem.

Mukbang has shown great potential in helping children with cancer to improve their appetite and food consumption, finally promote nutritional health. What's more, the features of Mukbang, such as high-quality and clear pictures, relaxed atmosphere created by the video makers, sounds while eating, and attractive images of food, may promote viewers' appetite and increase their intake imperceptibly. In addition to that, watching Mukbang while eating can also provide a pleasant eating experience for children with cancer, and the interaction with the Mukbang anchor can also alleviate the loneliness of children who live in hospital for such a long time, so as to enhance the children's taste experience, relieve the negative emotions of loneliness and depression.

Research has found that Mukbang can help people with low appetites increase their food intake and the interest in food. Several studies have shown that videos containing food cues can increase viewers' appetite and decrease feelings of satiety to a certain extent. At the same time, Mukbang can also increase viewers' taste experience on the basis of physics and improve children's interest in food. Thus, Mukbang is a useful tool for those who are struggling to increase the amount and variety of acceptable foods and gain weight. It also suggests that clinicians who treat eating disorders should be aware that Mukbang is a potential factor in their illness, and that effective positive use may be helpful for patients with anorexia or restrictive eating.

Given that, Mukbang will be applied to help children with cancer to improve appetite, nutritional status and quality of life. Studies have found that food images, eating sounds and interactivity of Mukbang may play a leading role in improving appetite. Thus, we defined the active ingredients of Mukbang as food images, eating sound and interactivity in this study. Based on that, this study aims to compare the effect of active ingredient Mukbang and general short videos without food cues on improving appetite in children with cancer, to provide evidence for larger randomized controlled trials (RCTS) and provide a new direction for clinical departments to develop nutritional interventions and management programs for children with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 6 to 18 years old;
* Children in accordance with the guidelines for the Diagnosis and Treatment of 12 Diseases related to hematologic diseases and malignant tumors (2021 version) issued by the General Office of the National Health Commission;
* At least experience one full cycle of chemotherapy;
* Children with moderate or higher symptoms of decreased appetite were screened for a list of treatment-related symptoms.

Exclusion Criteria:

* Children with serious cardiopulmonary disease, infection, organ damage, or genetic metabolic disease, immune deficiency disease, mental illness;
* Children with eye or ear dysfunction that prevents them from watching and listening to videos.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Self-reported appetite during the intervention | Change from baseline appetite during 7 days intervention
  A subjective sensation that stimulates the intake of food to provide the energy necessary for the most basic activities of life, which can be measured by the Cancer Appetite and Symptom Questionnaire (CASQ).
Self-reported appetite during the intervention | Change from baseline appetite at 4 weeks follow-up
  A subjective sensation that stimulates the intake of food to provide the energy necessary for the most basic activities of life, which can be measured by the Cancer Appetite and Symptom Questionnaire (CASQ).

SECONDARY OUTCOMES:
The level of nutritional status | Change from baseline nutritional status at 7 days
  Insufficient or excessive nutrient intake, imbalance of essential nutrients or impaired nutrient utilization, mainly manifested by wasting, stunting, underweight and micronutrient deficiency. Malnutrition is measured by the Subjective Global Nutritional Risk Assessment (SGNA).
The level of nutritional status | Change from baseline nutritional status at 4-weeks follow-up
  Insufficient or excessive nutrient intake, imbalance of essential nutrients or impaired nutrient utilization, mainly manifested by wasting, stunting, underweight and micronutrient deficiency. Malnutrition is measured by the Subjective Global Nutritional Risk Assessment (SGNA).
The level of the body mass index of the children with cancer | Change from baseline BMI at 7 days
  Body mass index (BMI), a simple method to evaluate the nutritional status and changes of children with cancer, which will be calculated as weight/height^2. Weight and height will be combined to report BMI in kg/m^2.
The level of the body mass index of the children with cancer | Change from baseline BMI at 4-weeks follow-up
  Body mass index (BMI), a simple method to evaluate the nutritional status and changes of children with cancer, which will be calculated as weight/height^2. Weight and height will be combined to report BMI in kg/m^2.
The quality of life after the intervention | Change from baseline quality of life at 7 days
  Individuals in different cultures and value systems experience their living conditions in relation to their goals, expectations, standards and concerns, including their physical health, mental state, independence, social relations, personal beliefs and relationships with the surrounding environment. This target is measured by the pediatric quality of life inventory measurement models 3.0 (PedsQLTM-3.0-cancer).
The quality of life after the intervention | Change from baseline quality of life at 4-weeks follow-up
  Individuals in different cultures and value systems experience their living conditions in relation to their goals, expectations, standards and concerns, including their physical health, mental state, independence, social relations, personal beliefs and relationships with the surrounding environment. This target is measured by the pediatric quality of life inventory measurement models 3.0 (PedsQLTM-3.0-cancer).

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The non-identified individual participant data will be shared after the outcomes have been published.
Supporting Information: SAP
Time Frame: After the publication of the study
Access Criteria: Researchers should contact the PI for approval of the study protocol.